CLINICAL TRIAL: NCT02481882
Title: Investigating Baseline Cortical Haemodynamics in Multiple Sclerosis
Brief Title: Baseline Cortical Haemodynamics in MS
Acronym: CortHaem
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15037
Record Dates: First submitted 2015-05-19; First posted 2015-06-25 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Magnetic Resonance Imaging; gadoteridol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Volunteers (Other): Healthy Volunteers will undergo an Magnetic Resonance Imaging scan.
  Interventions: Device: Magnetic Resonance Imaging
- MS Patients (Other): Patients will undergo and Magnetic Resonance Imaging scan including the use of Prohance (Gadoteridol).
  Interventions: Device: Magnetic Resonance Imaging; Drug: Prohance (Gadoteridol)

INTERVENTIONS:
Device: Magnetic Resonance Imaging — All scanning will be performed using a 7 Tesla Philips Achieva scanner with multi-transit capability (Philips Medical Systems, Best, The Netherlands). The volunteers will be scanned with a 32-channel receive coil.
Drug: Prohance (Gadoteridol) — A gadolinium based liquid administered intravenously in order to quantify blood flow in the brain using an MR scanner.
  Arms: MS Patients

SUMMARY:
This study will provide information on cortical haemodynamics in MS patients to address the discrepancies reported in previous literature, allowing further insight into the role of haemodynamics in the disease. It will also instruct us as to the most effective scanning protocols for future research. Developing a suitable protocol for studying perfusion longitudinally may also enable identification of new therapeutic interventions to normalise any perfusion abnormalities in MS patients.

DETAILED DESCRIPTION:
We aim to characterise the underlying cortical haemodynamics in Multiple Sclerosis (MS). We will assess two techniques for measuring blood flow in the brain: arterial spin labelling (ASL) and dynamic susceptibility contrast (DSC) magnetic resonance imaging in the MS patient group. ASL is a non-invasive technique whilst DSC-MR requires the administration of a tracer intravenously. Previous studies have shown conflicting results from these measurements. Reproducibility of ASL and disease activity will also be assessed through repeated scan sessions. Global perfusion in the MS patient group will be compared to a matched healthy control group.

In addition to measuring blood flow using both methods, we will investigate whether differences in perfusion between the MS patient group and the healthy controls can be observed using ASL, and also assess the reproducibility of ASL measurements via repeated scans. These repeated scanning sessions also provide a window to study disease activity in the patient cohort, and patients may be invited to return for up to a total of 4 scanning sessions (with only one involving the use of DSC) to better assess the usefulness of ASL in tracking haemodynamic changes in MS.

Study Regimen:

We aim to recruit 20 MS patients and 20 healthy age-matched controls for this study.

MS Patient Cohort:

The patients will be asked to attend two initial scanning sessions. MS Scan Session 1 will involve the use of the Prohance contrast agent, taking of blood samples and an MRI scan. MS Scan Session 2 will only involve the use of a non-invasive MRI scan.

MS Scan Session 1:

This session will require the administration of a gadolinium contrast agent. Prior to entering the scanner, a cannula is inserted into the patient's arm (cannula A). A small blood sample (5ml) will be taken from all MS patients in order to assess the haematocrit and creatinine content which will be used to determine if they are eligible for gadolinium administration (via use of the POCT i-Stat). This will provide a measure of eGFR which will provide information on the patient's renal function. This will only be performed once per patient and results will be recorded in the CRF. Provided the patient's eGFR is adequate for the study, a second cannula will be inserted into the patient's other arm (cannula B). The patient will enter the scanner with lines attached to both cannulae. The gadolinium bolus will be administered by a clinician in the scan room between scans via cannula A*. During the remainder of the visit, three subsequent blood samples will be taken (up to 5ml each), via cannula B, which will be used to measure gadolinium concentration. Gadolinium administration and blood work will be performed by physicians who are part of the research team with ALS training.

* Gadolinium contrast agents allow for the accurate quantification of blood flow from MR imaging. Prohance (Gadoteridol) is a gadolinium-based fluid administered intravenously to the participant. The contrast agent will be administered by physician with advanced life support (ALS) training. The physician will remain present throughout the duration of the scan and at all times whilst the participant is present at the Sir Peter Mansfield Imaging Centre. In the event of an emergency, a resuscitation kit is readily available. Also, the University's internal emergency phone number is contacted to readily direct emergency services to the site.

MS Scan Session 2:

The patients will be asked to return for MS Scan Session 2 two weeks after completing MS Scan Session 1. Before each scanning session, the patient will be asked to complete and MR safety questionnaire to ensure that no contraindications have arisen between scans. Explanations of what to expect in the MRI scanner environment will be given prior to being asked to sign a consent form. Provided there are no contraindications for the volunteer to enter the scanner, the volunteer will undergo a non-invasive MRI scan lasting approximately 1 hour. No other interventions are to be used. All scanning will be performed using a 7 Tesla Philips Achieva scanner with multi-transit capability (Philips Medical Systems, Best, The Netherlands). The participants will be scanned with a 32-channel receive coil. The subjects will wear-ear plugs, ear defenders and a pulse oximeter (to monitor the pulse) throughout contrast agent administration.

After the completion of MS Scan Sessions 1 and 2, their scans will be analysed and interpreted by a member of the patient's clinical care team. If a patient presents any morphological changes relating to the disease between MS Scan Sessions 1 and 2, the patient will be invited back for an additional 2 scans, labelled as MS Scan Session 3 and 4. If there is no presentation of additional lesions between scans, this will be the end of the patient's participation.

MS Scan Sessions 3 and 4:

These will be identical to MS Scan Session 2 (non-invasive MRI scan only). MS Scan Session 3 will take place at 6 weeks and MS Scan Session 4 will take place at 12 weeks.

Healthy Volunteers:

The healthy volunteers will be asked to attend two scanning sessions (labelled as HV Scan Session 1 and HV Scan Session 2 in the flow chart). Both HV Scan Session 1 and 2 will only involve the use of a non-invasive MRI scan. No gadolinium contrast agent is to be given to the healthy volunteers during this study.

Both HV Scan Session 1 and 2 will be identical to MS Scan Sessions 2, 3 and 4. Upon completing HV Scan Session 1, the healthy volunteer will be invited back for HV Scan Session 2 two weeks later. After completing HV Scan Session 2, the healthy volunteer's participation will be finished.

ELIGIBILITY:
Inclusion Criteria (Healthy Volunteers):

* Male or female volunteers who are between the ages of 21 and 80.
* Able to give voluntary written informed consent to participate in the study.
* Able to understand the requirements of the study, including anonymous publication, and agree to co-operate with the study procedures.

Inclusion Criteria (Patients):

* Diagnosed with Multiple Sclerosis.
* Male or female volunteers who are between the ages of 21 and 80.
* Able to give voluntary written informed consent to participate in the study.
* Able to understand the requirements of the study, including anonymous publication, and agree to co-operate with the study procedures.

Exclusion Criteria:

* Any history of neurological illness other than MS.
* Known hypersensitivity to any MR or X-Ray contrast agent.
* Any history of renal failure or disease.
* Any history of allergies.
* Any history of circulation problems (vascular disease).
* Pregnancy or breastfeeding.
* MRI contraindications as screened on safety questionnaire (e.g. metal implants or pacemaker).
* Have taken part in any other clinical study within the previous 3 months.#
* Any contraindications provided from MRI or contrast agent safety forms.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Cerebral Blood Flow | 1 hour
  A short MRI scan is able to quantify the amount of blood perfusion into brain tissue (to be performed with and without the gadolinium contrast agent).

SECONDARY OUTCOMES:
Arterial Cerebral Blood Volume | 1 hour
  A short MRI scan is able to quantify the volume of arterial blood in a volume of brain tissue.
Arterial Transit Time | 1 hour
  A short MRI scan is able to quantify the amount of time taken for blood to reach an area of the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Evangelou, Ph.D., Principal Investigator — Faculty of Medicine & Health Sciences
Locations (1):
- Queen's Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No